CLINICAL TRIAL: NCT06023862
Title: A Three-arm Randomized Phase II Study of Dostarlimab Alone or With Bevacizumab Versus Nonplatinum Chemotherapy in Recurrent Gynecological Clear Cell Carcinoma: DOVE (APGOT-OV07/ ENGOT-ov80 Study)
Brief Title: A Three-arm Randomized Phase II Study of Dostarlimab Alone or With Bevacizumab Versus Nonplatinum Chemotherapy in Recurrent Gynecological Clear Cell Carcinoma: DOVE (APGOT-OV7/ ENGOT-ov80 Study)
Acronym: DOVE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, JUNGYUN LEE, Professor, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2023-0794
Record Dates: First submitted 2023-08-23; First posted 2023-09-05 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Ovarian Neoplasms; Endometrial Neoplasms; Uterine Cervical Neoplasms; Vulvar Cancer; Vagina Neoplasm; Clear Cell Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms; Uterine Cervical Neoplasms; Vulvar Neoplasms; Vaginal Neoplasms; Adenocarcinoma, Clear Cell | interventions — dostarlimab; Bevacizumab; Doxorubicin; Gemcitabine; Paclitaxel; liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (Experimental): Dostarlimab monotherapy
  Interventions: Drug: Dostarlimab
- Group B (Experimental): Dostarlimab + Bevacizumab combination therapy
  Interventions: Drug: Dostarlimab; Drug: Bevacizumab
- Group C (Active Comparator): General chemotherapy (one of Pegylated liposomal doxorubicin, Doxorubicin, Paclitaxel, and Gemcitabine)
  Interventions: Drug: Doxorubicin; Drug: Gemcitabine; Drug: Paclitaxel; Drug: Pegylated liposomal doxorubicin

INTERVENTIONS:
Drug: Dostarlimab — Intravenous (IV) infusion
  Other Names: Jemperli
  Arms: Group A; Group B
Drug: Bevacizumab — Intravenous (IV) infusion
  Arms: Group B
Drug: Doxorubicin — Intravenous (IV) infusion
  Arms: Group C
Drug: Gemcitabine — Intravenous (IV) infusion
  Arms: Group C
Drug: Paclitaxel — Intravenous (IV) infusion
  Arms: Group C
Drug: Pegylated liposomal doxorubicin — Intravenous (IV) infusion
  Arms: Group C

SUMMARY:
Multicenter, randomized, open-label, phase II clinical study comparing Dostarlimab +/- Bevacizumab with standard chemotherapy in patients with gynecological clear cell carcinoma.

198 subjects will be enrolled in this study and will be assigned to three groups in a 1:1:1 ratio.

1. Group A: Dostarlimab monotherapy

   * First 3 cycles: Dostalimab 500mg every 3 weeks, IV
   * 4 cycles ~ up to 24 months: Dostalimab 1000mg every 6 weeks, IV
2. Group B: Dostarlimab + Bevacizumab combination therapy

   * First 3 cycles: Dostalimab 500mg every 3 weeks, IV
   * 4 cycles ~ up to 24 months: Dostalimab 1000mg every 6 weeks, IV
   * Bevacizumab administered IV at 15 mg/kg every 3 weeks until disease progression or unacceptable toxicity
3. Group C: General chemotherapy (one of Pegylated liposomal doxorubicin, Doxorubicin, Paclitaxel, and Gemcitabine)

ELIGIBILITY:
Inclusion Criteria:

1. Female patient is at least 18 years of age,
2. Patient has signed the Informed Consent (ICF) and is able to comply with protocol requirements.
3. Patient with histologically proven confirmed recurrent or persistent clear cell carcinoma of the ovary, endometrium, cervix, vagina, and vulva

   * Local review by gynecologic pathologist required
   * ≥50% clear cell histology in case of mixed carcinoma
   * WT-1 neg (Only in case of ovarian cancer) Note: In the case of including non-ovarian clear cell carcinoma with more than 20 cases, the decision is made through discussion with the SPONSOR.
4. Patient with an Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
5. Disease progression within 12 months of completing platinum-based chemotherapy
6. 1-5 prior lines of therapies
7. Patient with measurable disease according RECIST 1.1 criteria
8. Availability of Tumor tissue for translational research . - A formalin-fixed paraffin-embedded (FFPE) tumor block(preferred) or at least 20 slides (unstained, freshly cut, serial sections) must be submitted.
9. Patients who consent to fresh tumor biopsies

   * Confirmed with at least one lesion with location accessible to safely biopsy per the clinical judgement of the investigator
   * Note: If mandatory biopsies cannot be performed as per investigator's clinical judgement, discussion and agreement between investigator and Sponsor are required.
10. Patient has adequate organ function, defined as follows:

    1. Absolute neutrophil count ≥ 1,500 cells/μL
    2. Platelets ≥ 100,000 cells/μL
    3. Hemoglobin ≥ 9 g/dL or ≥ 5.6 mmol/L
    4. Serum creatinine ≤ 1.5× upper limit of normal (ULN) or calculated creatinine clearance ≥ 50 mL/min using the Cockcroft-Gault equation for patients with creatinine levels > 1.5× institutional ULN
    5. Total bilirubin ≤ 1.5× ULN (≤ 2.0 x ULN in patients with known Gilbert's syndrome) or direct bilirubin ≤ 1× ULN
    6. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5× ULN unless liver metastases are present, in which case they must be ≤ 5× ULN
    7. International normalized ratio or prothrombin time (PT) ≤1.5× ULN and activated partial thromboplastin time ≤1.5× ULN.Participants taking anticoagulants may be included on a stable dose with a therapeutic INR <3.5. .
11. Patient must have a negative serum pregnancy test within 72 hours of the first dose of study medication, unless they are of non-childbearing potential. If a negative result cannot be confirmed by a urine test, a serum pregnancy test is required. Non-childbearing potential is defined as follows:

    1. Patient is ≥ 45 years of age and has not had menses for > 1 year.
    2. A follicle-stimulating hormone value in the postmenopausal range upon screening evaluation if amenorrhoeic for < 2 years without a hysterectomy and oophorectomy.
    3. Post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation:

       * Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound, MRI, or CT scan.
       * Tubal ligation must be confirmed with medical records of the actual procedure.
       * Information must be captured appropriately within the site's source documents.
12. Patient of childbearing potential must agree to use a highly effective method of contraception with their partners starting from time of consent through 180 days after the last dose of study treatment. Note: Abstinence is acceptable if this is the established and preferred contraception for the patient (Information must be captured appropriately within the site's source documents).

Exclusion Criteria:

1. Patient has had ≥ 6 prior lines of chemotherapy. Surgery of the recurrence is allowed.
2. Patient has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
3. Patient has received prior anticancer therapy (chemotherapy, targeted therapies, hormonal therapy, radiotherapy) within 21 days or < 5 times the half-life of the most recent therapy prior to Study Day 1, whichever is shorter.

   Note: Palliative radiation therapy to a small field ≥ 1 week prior to Day 1 of study treatment may be allowed after discussion with the SPONSOR.
4. Patient with contraindication to chemotherapy or immune checkpoint inhibitor treatments or anti-angiogenic inhibitor
5. Patients with uncontrolled hypertension (defined as systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥100 mmHg) based on an average of ≥ 3 BP readings on ≥ 2 sessions.
6. Patients with evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
7. Patients with current abdominal/pelvic fistula
8. Patient has a concomitant malignancy, or patient has a prior non-gynecological malignancy who has been disease-free for < 3 years or who received any active treatment in the last 3 years for that malignancy. Non-melanoma skin cancer is allowed.
9. Patient has known uncontrolled central nervous system metastases, carcinomatosis meningitis, or both. Note: Patients with previously treated brain metastases may participate provided they are stable (without evidence of disease progression by imaging [using the identical imaging modality for each assessment, either MRI or CT scan] for at least 4 weeks prior to the first dose of study treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and have not been using steroids for at least 7 days prior to study treatment. Carcinomatous meningitis precludes a patient from study participation regardless of clinical stability.
10. Patient has a known history of human immunodeficiency virus (HIV; HIV ½ antibodies). Participants with known human immunodeficiency virus(HIV) are allowed if they meet all of the following criteria:

    * Cluster of differentiation 4(CD4) ≥350/μL and viral load <50 copies/mL.
    * No history of acquired immunodeficiency syndrome-defining opportunistic infections within 12 months before enrollment.
    * No history of HIV-associated malignancy for the past 5 years.
    * Concurrent antiretroviral therapy as per the most current National Institutes of Health (NIH) Guidelines for the Use of Antiretroviral Agents in Adults and Adolescents with HIV started >4 weeks before study enrollment.
11. Patient with presence of hepatitis B surface antigen or a positive hepatitis C antibody test result at screening or within 3 months before first dose of dostarlimab treatment.

    * Participants who are hepatitis B surface antigen positive may be enrolled if their HBV-DNA level is below the institutional lower limit.
    * Participants with chronic hepatitis B virus (HBV) infection who meet the criteria for anti-HBV therapy may be eligible if the participant is on a suppressive antiviral therapy before initiation of cancer therapy.
    * Participants with positive hepatitis C antibody due to prior resolved disease can be enrolled only if a confirmatory negative hepatitis C RNA polymerase chain reaction is obtained. Hepatitis C participants may be eligible if they both have completed curative therapy and have a hepatitis C viral load <!-- Not Allowed Tag Filtered --><quantifiable limit.
12. Patient has an active autoimmune disease that required systemic treatment in the past 2 years. Replacement therapy is not considered a form of (eg, thyroid hormone or insulin).
13. diagnosis immunodeficiency receiving steroid any other immunosuppressive within 7 days prior to first dose study treatment. Patients who have received acute and>/or low-dose systemic immunosuppressive medications (e.g,, a one-time dose of dexamethasone for nausea or chronic use of ≤ 10 mg/day of prednisone or dose equivalent corticosteroid) may be enrolled in the study after discussion with and approval by the Sponsor. The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) is allowed.
14. Patient has not recovered (to Grade ≤ 1) from previous anti-cancer therapy-induced adverse events (AEs).

    Note: Patients with Grade ≤ 2 neuropathy, Grade ≤ 2 alopecia, or Grade ≤ 2 fatigue are an exception to this criterion and may qualify for the study.
15. Patient has not recovered adequately from AEs or complications from any major surgery prior to starting therapy. Major surgical procedures, other than for diagnosis, within 4 weeks prior to initiation of study treatment
16. Patient has a known hypersensitivity to bevacizumab or dostarlimab components or excipients.
17. Patient is currently participating and receiving study treatment or has participated in a study of an investigational agent and received study treatment or used an investigational device within 4 weeks of the first dose of treatment.
18. Patient is considered a poor medical condition due to a serious, uncontrolled medical disorder, non-malignant systemic disease, or active infection requiring systemic therapy. Specific examples include, but are not limited to, active, non-infectious pneumonitis; uncontrolled ventricular arrhythmia; recent (within 90 days) myocardial infarction; uncontrolled major seizure disorder; unstable spinal cord compression; superior vena cava syndrome; or any psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study (including obtaining informed consent).
19. Patients with known history of non-infectious pneumonitis that required steroids or has current pneumonitis.
20. Use of any of the following immunomodulatory agents within 28 days prior to the first dose of study drug:

    * Interferons
    * Interleukins
    * Live vaccine Note: Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster, yellow fever, rabies, BCG, and typhoid vaccine. mRNA and adenoviral-based COVID-19 vaccines are considered non-live and are not exclusionary. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed as other killed vaccines, if done at least 2 weeks prior the first dose of study drug; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
21. Patient who are pregnant or lactating, or plan to become pregnant or lactate during the expected duration of the study, from screening through 180 days after the last dose of study drug.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | Up to approximately 48 months
  The time from the date of randomization until first documentation of disease progression, as determined by investigator assessment based on RECIST 1.1, or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Objective Response Rate | Up to approximately 48 months
  the proportion of patients who have best overall response of either complete response (CR) or partial response (PR), as investigator assessment based on RECIST 1.1
Disease control rate | Up to approximately 48 months
  the proportion of patients who have best overall response of CR, PR, or stable disease (SD) by investigator assessment per RECIST 1.1 . SD must be achieved at ≥ 7 weeks after randomization to be considered best overall response.
Clinical benefit rate | Up to approximately 48 months
  the proportion of patients who have best overall response of CR, PR, or stable disease (SD) by investigator assessment per RECIST 1.1 . (duration of SD ≥ 23 weeks after randomization)
Progression Free Survival 2 | Up to approximately 72 months
  the time from initial randomization to the second objective disease progression (ie, after the first subsequent therapy) or death.
Overall survival | Up to approximately 72 months
  the time from the date of randomization until death due to any cause
Duration of Response Rate | Up to approximately 48 months
  Measured from the time of initial response until documented tumor progression.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Up to approximately 72 months
  Assessed by CTCAE v5.0 (by investigators).
Time to first and second Subsequent Treatment | Up to approximately 72 months
  the time from the date of randomization to date of the first and second subsequent anticancer therapy or death.
Response rate of subsequent therapies | Up to approximately 72 months
  the proportion of patients who have best overall response of either complete response (CR) or partial response (PR), as investigator assessment based on RECIST 1.1

OTHER OUTCOMES:
Disease-related or Treatment-related Biomarkers | At the end of study, Up to approximately 72 months
  Translational research including NGS as well as MMRd, MSI-H, PD1/L1, TMB, Immune signature, and Tie-2.
Comparison of RECIST1.1 and i-RECIST assessment | Throughout duration of study, Up to 48 months
  By comparing RECIST 1.1 and iRECIST, evaluate the accuracy of iRECIST for assessing the therapeutic efficacy of ICIs.

CONTACTS AND LOCATIONS:
Overall Officials: JUNGYUN LEE, Ph.D., Principal Investigator — Severance Hospital, Yonsei University Health System
Locations (18):
- Japan (10):
  - Kurume University Hospital, Kurume, Fukuoka
  - Fukushima Medical University Hospital, Fukushima, Fukushima
  - Mie University Hospital, Tsu, Mie-ken
  - Tohoku University Hospital, Sendai, Miyagi
  - Niigata Cancer Center Hospital, Niigata, Niigata
  - Saitama Medical University International Medical Center, Hidaka, Saitama
  - Tokushima University Hospital, Tokushima, Tokushima
  - The Jikei University Hospital, Tokyo, Tokyo
  - The Cancer Institute Hospital Of JFCR, Tokyo, Tokyo
  - University of Tsukuba Hospital, Tsukuba, ㅊ Ibaraki
- National University Hospital, Singapore, Singapore
- South Korea (7):
  - Severance Hospital, Yonsei Health System, Seoul, Seoul
  - National Cancer Center, Goyang-si
  - Bundang Seoul National University Hospital, Seongnam-si
  - Asan Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University, Seoul

REFERENCES:
- [Derived] Lee JY, Tan D, Ray-Coquard I, Lee JB, Kim BG, Van Nieuwenhuysen E, Huang RY, Tse KY, Gonzalez-Martin A, Scott C, Hasegawa K, Wilkinson K, Yang EY, Lheureux S, Kristeleit R. Phase II randomized study of dostarlimab alone or with bevacizumab versus non-platinum chemotherapy in recurrent gynecological clear cell carcinoma (DOVE/APGOT-OV7/ENGOT-ov80). J Gynecol Oncol. 2025 Jan;36(1):e51. doi: 10.3802/jgo.2025.36.e51. Epub 2024 Dec 16. PMID 39710508